CLINICAL TRIAL: NCT05444179
Title: The Effectiveness of Nutrition and Physical Activity Intervention on Psychosocial Well-Being of Mothers With Preterm Infants in Selangor
Brief Title: Nutrition and Physical Activity Intervention on Psychosocial Well-Being of Postpartum Mothers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Teknologi Mara (Other)
Collaborators: Universiti Sains Islam Malaysia (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Nur Islami Bt Mohd Fahmi Teng, Assoc. Prof/ Principle Investigator, Universiti Teknologi Mara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MiChild Group
Record Dates: First submitted 2022-04-13; First posted 2022-07-05 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Postpartum Depression; Lifestyle, Healthy
Keywords: postpartum depression; physical activity; intervention study; nutritional intake
MeSH Terms: conditions — Depression, Postpartum; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group study design, which employed block randomization via a computer-generated randomisation list for allocation of the participants, with the block size of 8, and equal randomization ratio (1:1) between intervention and control groups. The block randomization process is conducted by an investigator that had no clinical involvement in the trial, in which the allocation sequence was concealed from the principal investigator who are enrolling and assessing the eligible participants. Due to nature of intervention, blinding of principal investigator and participants are not possible. Measurement of the outcome will commence at the baseline, at week 4 and week 8 of the randomised controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): The participant will be provided an educational module entitled "Mommies can Eat and Exercise with No Stress" (MomEENS), in which the module will be delivered through a booklet and video. The MomEENS module consist of five key recommendations: 1. Eat healthy foods ;2. Eat foods rich in iron and folic acid; 3. Eat foods rich in omega-3 fatty acids; 4. Increase steps in a day and; 5. Increase body flexibility and strength. All the key recommendations will be explained in the booklet, while the video will provide full guidance on how to exercise during postpartum at home, explaining key recommendations 4 and 5. Face-to-face consultation with the participants will be held during baseline and 4th week to enhance the participation. Besides, Whatsapp and Facebook page group is developed as a step to enhance the compliance of participants. All the participants will be contacted once for every two weeks, lasting for about 5 to 10 minutes for each call to monitor the participant's progress.
  Interventions: Behavioral: Mommies can Eat & Exercise with No Stress (MomEENS)
- Control group (No Intervention): The participants in the control group will be received advice on the standardised Malaysian food pyramid and be instructed to follow their usual standard care as suggested by their healthcare provider. Postpartum women in Malaysia typically attend postpartum healthcare visits with an exam on day 30 after childbirth but receive no other routine care following this appointment unless a specific health problem has been identified. Participants in the control group performed the same evaluations. They received the same incentives as those in the intervention group, but they did not receive any educational module and contact from the investigator during the 8 weeks follow-up.

INTERVENTIONS:
Behavioral: Mommies can Eat & Exercise with No Stress (MomEENS) — This intervention involving behaviour modification, incorporates nutrition and physical activity modification. The intervention encourages participants to consume a healthy diet and active lifestyle during postpartum period. For nutrition modification, a general advice on healthy nutrition were given and several nutrients are highlighted which evidenced can reduce postpartum depression. While for physical activity, the mothers are encouraged to do exercise, targeting aerobic, flexibility, and strength type of exercise. The exercise protocol is progressive. During the first month, the participants will be advised to conduct flexibility and strength exercises for 8 repetitions (1 set), at least 3 days per week for both aerobic and flexibility exercise. While during the second month, participants are asked to increase repetitions and frequency of exercises, up to 16 repetitions (2 set) for each flexibility exercise, and conduct exercise at least 5 days per week.
  Arms: Intervention group

SUMMARY:
This study aims to examine the effectiveness of nutrition and physical intervention to improve psychosocial well-being of postpartum mothers with preterm infants. The focus was highlighted towards the mothers of preterm infants who were cared in Neonatal Intensive Care Unit (NICU) as these parents might have a higher stress level than the full-term infants. The intervention consisted of a module designed for postpartum mothers, incorporating nutrition and physical activity entitled Mommies can Eat & Exercise with No Stress (MomEENS).

DETAILED DESCRIPTION:
The intervention is aim to encourage the participant to have better nutrition intake and engage in low to moderate-intensity exercise on 3 to 5 days per week, for 8 weeks in order to improve their psychosocial well-being. After being informed about the study and potential risks, the participants will be screened according to their eligibility criteria. The participants who are eligible to participate in the study will be contacted again and asked for consent to join the study. After obtaining the consent, the participant will undergo a baseline assessment, and subsequently, the investigator will assign the participant to their respective groups, the intervention and control groups. All of the health assessments will be conducted at baseline, 4th week and 8th week.

In intervention group, the participant will be provided an educational module entitled "Mommies can Eat and Exercise with No Stress" (MomEENS), in which the module will be delivered through a booklet and video. The MomEENS module incorporated achievement-based objectives for five key recommendations: 1. Eat healthy foods ;2. Eat foods rich in iron and folic acid; 3. Eat foods rich in omega-3 fatty acids; 4. Increase steps in a day and; 5. Increase body flexibility and strength. All the key recommendations will be explained in the booklet, while the video will provide full guidance on how to exercise during postpartum at home, explaining key recommendations 4 and 5.

Face-to-face consultation with the participants will be held at baseline and 4th week to enhance the participation and motivation of the participants towards the intervention. Besides, Whatsapp and Facebook page group is developed as a step to enhance the compliance of participants towards intervention. The group will be created soon after the participants undergo the baseline phase. Whatsapp group provides a medium for participant to ask, share, and communicate with other participants (only within the intervention group) regarding the intervention activities they commit. On the other hand, Facebook page group will provide a forum to support and additional related information. In addition to the continuity of the compliance, telephone follow-up calls will be at least administered once for every two weeks, lasting for about 5 to 10 minutes for each call. It is aimed to monitor the participant's progress while engaging in appropriating self-management behaviours.

The participants in the control group will be received advice on the standardised Malaysian food pyramid and be instructed to follow their usual standard care as suggested by their healthcare provider. Postpartum women in Malaysia typically attend postpartum healthcare visits with an exam on day 30 after childbirth but receive no other routine care following this appointment unless a specific health problem has been identified. Participants in the control group performed the same evaluations. They received the same incentives as those in the intervention group, but they did not receive any educational module and contact from the investigator during the 8 weeks follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with EPDS score ≥ 12
2. Mothers with an infant nearly graduated from NICU due to prematurity with minimum stays of 7 days (Gestational age: < 37 weeks).
3. Postpartum mothers (within 4th to 8th weeks after childbirth).
4. Aged between 19 until 40 years old.
5. Mothers were from Malaysian citizen.
6. Mothers who only reside in Selangor, Klang Valley or Negeri Sembilan during their postpartum confinement.
7. Only Malay mothers will be selected (due to small number population on Chinese and Indian, following from Phase 1)
8. Mothers who undergo vaginal delivery for the current child.
9. Mothers who are fit to do exercise, based on the 10-item Physical Activity Readiness Questionnaire (PAR-Q).

Exclusion Criteria:

1. Mothers that is clinically diagnosed with mental illness or other known psychiatric disorders
2. Mothers who illiterate either in Malay or English
3. Mothers who are currently pregnant
4. Mothers whose infant has genetic or congenital anomaly or severe cardiorespiratory instability
5. Mothers who have chronic or terminal disease (such as cancer, renal failure, hypothyroid, exercised-induced asthma and uncontrolled hypertension and diabetes) or diseases that would limit to exercise.
6. Mothers who have any condition that would make exercise unsafe or unwise.

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only postpartum female is eligible in this study
Enrollment: 32 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale | Change from Baseline Depression Screening Status at 8 weeks
  The presence of depressive symptoms will be assessed using the Edinburgh Postnatal Depression Scale (EPDS). The EPDS is a 10-item self-administered questionnaire designed specifically to measure postpartum depression. All items will be rated on a 4-point Likert-type scale, with a total score ranging from 0-30. Categories of response are scored 0,1,2, and 3 based on increased symptom severity. EPDS can only be used for screening but not for the clinical diagnosis of depression. The Malay version of the scale was validated in the local setting with the cut off 11/12 was used to determine a woman at risk of having depressive symptoms. Score of ≥12 indicates the presence of postpartum depression whereas <12 indicates absence of postpartum depression.
Perceived Stress Scale (PSS) | Change from Baseline Perceived Stress Status at 8 weeks
  The Perceived Stress Scale (PSS) was developed by Sheldon Cohen & Williamson (1988), designed to measure the degree to which circumstances of an individual are considered stressful via their feelings and thoughts in the past month. The item asked regarding the current levels of stress, unpredictable, uncontrollable, and overloaded events, unexpectedly occur during their lives. The PSS consist of 10 items, derived from 5-point Likert scale (0= never, 1= almost never, 2= sometimes, 3= fairly often, 4= very often). Four items that are positively stated (item 4,5,7, and 8) are scored reversely (0= very often, 1= fairy often, 2= sometimes, 3= almost never, 4= never). The total score is calculated from the sum of 10 items, whereas higher scores indicate higher levels of perceived stress. In this study, Malay version of PSS-10 is used to enable participants to understand the questions asked and to make the assessment more culturally appropriate.
Postpartum Sleep Quality Scale (PSQS) | Change from Baseline Sleep Quality Status at 8 weeks
  The Postpartum Sleep Quality Scale (PSQS) consists of 14 item scale, designed to assess subjective sleep quality during postpartum periods. Two domains were developed from the PSQS: "Factor 1: Infant night care-related daytime dysfunction", and "Factor 2: Physical symptoms related sleep inefficiency". Factor 1 explained how having care of infants at night impacted the quality of postpartum woman's sleep and the ability to handle daytime activities. Factor 2 described the physiological factors underlying sleep and sleep inefficiency symptoms of a woman. The PSQS found to be a valid and reliable tool, as previous study had demonstrated PSQS have adequate internal consistency between the item (Cronbach's α= 0.88; Factor I α =0.89, Factor II α= 0.82).
Positive Affect Balance Scale (PABS) | Change from Baseline Psychosocial Well-being Status at 8 weeks
  This scale consist of 10 item scales, which 5 items were developed for each positive and negative affect components, asking the psychological reactions of people respond to their daily lives, and individual's ability to cope with daily stresses. "Positive affect" questions are associate to social participation, satisfaction with social life, and engagement in activities. Three-point scale of "never", "sometimes", or "often" are answers made to the questions represents the past week's experiences. All calculations of positive affect score, a negative affect score and a total affect balance score can be made. The positive impact score (ranging from 5 to 15) with 15 being the highest (most positive result) will be used in this study. PABS has been proven to be a reliable tool for measuring psychosocial well-being, as reported by previous study.

SECONDARY OUTCOMES:
Multiple Pass 24-Hour Diet Recall | Change from Baseline Dietary Intake at 8 weeks
  A multiple pass 24-hour diet recall will be performed to assess the dietary intake of the mother. Multiple pass 24-hour diet recall found to maximise recall accuracy for quantitation, with the used of the following algorithm: The first pass encourages the respondent to freely report all food and drink consumption for the previous 24 hours without any interruption. In second pass, the researcher probes for greater details on the exact time, type and quantity of food and drink consumed, and in the final pass, the researcher reviews all food reported in order, prompting for omissions and clarifying the ambiguities. Nutrient analysis software, the Nutritionist Pro Diet Analysis, will be used to calculate the average nutrients intake, which is based on the Nutrient Composition of Malaysian Foods database and the U.S. Department of Agriculture (USDA) Foods database.
International Physical Activity Questionnaire- Short Form | Change from Baseline Physical Activity Status at 8 weeks
  This is a self-report questionnaire that assesses the types of intensity of physical activity and sitting time that people do as part of their daily lives. are considered to estimate total physical activity in MET-min/week and time spent sitting. There are 7 items asking for the number of days a week they participated in the activities and the average time for each session on each activity (hours and minutes) they spent during the past 7 days. The intensity score is then calculated based on the MET classification levels (low, moderate, high).
Body weight measurement | Change from Baseline Body Weight at 8 weeks
  Weight is measured to the nearest 0.1 kilogram (kg) with a portable standard scale using Seca 813 Electronic Flat (Birmingham, United Kingdom) weighing scale.
Height measurement | Change from Baseline Height Measurement at 8 weeks
  Height of the participant is measured to the nearest 0.1cm using Seca 217 Height Measure (Birmingham, United Kingdom).
Waist circumference measurement | Change from Baseline Waist Circumference at 8 weeks
  Waist circumference is measured to the nearest 0.1cm using Seca 201 Ergonomic circumference measuring tape (Birmingham, United Kingdom).
Blood Pressure Assessment | Change from Baseline Blood Pressure Assessment at 8 weeks
  Systolic and diastolic blood pressure is measured using automated non-invasive blood pressure monitor device with cuff, Omron Blood Pressure Monitor HEM 7120 (Kyoto, Japan).
Breastfeeding Self-Efficacy -Short Form (BSES-SF) | Change from Baseline Breastfeeding Self-Efficacy at 8 weeks
  The Breastfeeding Self-Efficacy Scale- Short Form (BSES-SF) is a self-report instrument developed to measure breastfeeding confidence. BSES-SF consist of 14 items, with each item is followed by the phrase "I can always". The answer option is assisted with a 5-point Likert-type scale where 1 indicates not at all confident and 5 indicates always confident. The sum of all items will be in the range of 14 for the minimum score, and 70 is the maximum score, which indicates the data as continuous. BSES-SF is a very excellent measure of breastfeeding efficacy as it has shown a high reliability (with Chronbach's Alpha value is 0.97) and validity score (BSES-SF is significantly correlated (p< 0.05) with other theoretically related concepts (self-esteem, postpartum depression and perceived stress).

CONTACTS AND LOCATIONS:
Overall Officials: Nur Islami Bt Mohd Fahmi Teng, AP. Dr., Principal Investigator — Universiti Teknologi Mara
Locations (1):
- Universiti Teknologi MARA, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arifin, S. R. M., Ahmad, A., Rahman, R. A., Loh, H. S., & Ng, C. G. (2014). Postpartum depression in Malaysian women: The ssociation with the timing of pregnancy and sense of personal control during childbirth. International Journal of Academic Research, 6(3), 143-149. https://doi.org/10.7813/2075-4124.2014/6-3/b.20
- [Background] Cohen, S., & Williamson, G. (1988). Perceived Stress in a Probability Sample of the United States. Sage.
- [Background] Dennis CL. The breastfeeding self-efficacy scale: psychometric assessment of the short form. J Obstet Gynecol Neonatal Nurs. 2003 Nov-Dec;32(6):734-44. doi: 10.1177/0884217503258459. PMID 14649593
- [Background] Husin, H., Isa, Z. M., Ariffin, R., Rahman, S. A., & Ghazi, H. F. (2017). The Malay version of antenatal and postnatal breastfeeding self-efficacy scale-short form: Reliability and validity assessment. Malaysian Journal of Public Health Medicine, 17(2), 62-69.
- [Background] Mahmud WM, Awang A, Mohamed MN. Revalidation of the Malay Version of the Edinburgh Postnatal Depression Scale (EPDS) Among Malay Postpartum Women Attending the Bakar Bata Health Center in Alor Setar, Kedah, North West Of Peninsular Malaysia. Malays J Med Sci. 2003 Jul;10(2):71-5. PMID 23386800
- [Background] Moriwaki SY. The affect balance scale: a validity study with aged samples. J Gerontol. 1974 Jan;29(1):73-8. doi: 10.1093/geronj/29.1.73. No abstract available. PMID 4809667
- [Background] Sandhu SS, Ismail NH, Rampal KG. The Malay Version of the Perceived Stress Scale (PSS)-10 is a Reliable and Valid Measure for Stress among Nurses in Malaysia. Malays J Med Sci. 2015 Nov;22(6):26-31. PMID 28223882
- [Background] Nightingale H, Walsh KJ, Olupot-Olupot P, Engoru C, Ssenyondo T, Nteziyaremye J, Amorut D, Nakuya M, Arimi M, Frost G, Maitland K. Validation of triple pass 24-hour dietary recall in Ugandan children by simultaneous weighed food assessment. BMC Nutr. 2016 Aug 24;2:56. doi: 10.1186/s40795-016-0092-4. PMID 27795836
- [Background] Yang CL, Chen CH. Effectiveness of aerobic gymnastic exercise on stress, fatigue, and sleep quality during postpartum: A pilot randomized controlled trial. Int J Nurs Stud. 2018 Jan;77:1-7. doi: 10.1016/j.ijnurstu.2017.09.009. Epub 2017 Sep 14. PMID 28950158
- [Background] Yang CL, Yu CH, Chen CH. Development and validation of the postpartum sleep quality scale. J Nurs Res. 2013 Jun;21(2):148-54. doi: 10.1097/jnr.0b013e3182921f80. PMID 23681351

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT05444179/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-21): https://cdn.clinicaltrials.gov/large-docs/79/NCT05444179/ICF_001.pdf